CLINICAL TRIAL: NCT00506818
Title: Cognitive and Emotional Impairment After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Asker og Baerum (Other)
Collaborators: University of Oslo (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1.2006.2076(REK); 1.2006.2076(REK); 16307(NSD)
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Last update posted 2009-09-21 (Estimated); Status verified 2009-09

CONDITIONS: Stroke; Cognitive Impairment; Vascular Dementia
Keywords: emotional symptoms; vascular risk-factors
MeSH Terms: conditions — Stroke; Cognitive Dysfunction; Dementia, Vascular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2 (Active Comparator): Intensive risk factor intervention
  Interventions: Other: Multifactorial vascular-risk-factor-intervention

INTERVENTIONS:
Other: Multifactorial vascular-risk-factor-intervention

SUMMARY:
Cognitive and emotional symptoms are often seen in the acute phase of a stroke. The prevalence of such symptoms later and the mechanisms explaining the symptoms are not fully known. The causes of poststroke dementia are likely to be multifactorial (Cerebrovascular Diseases 2006). The investigators want to include all patients with first ever stroke without significant cognitive decline prior to the stroke (IQCODE cut-off 3,7) and follow them up for one year. At baseline we will make stroke classifications, measure neurological deficits according to NIHSS, evaluate cognitive and emotional function and make registrations of vascular risk factors, including precerebral color duplex scan with measurement of IMT in CCA. The investigators will then randomize the patients into multifactorial vascular-risk-factor-intervention in the hospital or care as usual in the primary health care. 8-12 months after stroke onset, survivors will undergo new examinations to evaluate neurological, cognitive and emotional functions, as well as MRI and SPECT.

ELIGIBILITY:
Inclusion Criteria:

* First ever stroke or TIA
* No cognitive decline (IQCODE < 3,7)
* Survived the acute stroke
* Expected to live at least for one year after stroke

Exclusion Criteria:

* Cognitive decline

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2007-02; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Effects of vascular risk-factor-intervention on changes in TMTA, ten-words-test and HAD | 8-12 months after stroke onset

SECONDARY OUTCOMES:
Prevalence of dementia and depression after stroke | 8-12 month after stroke onset

CONTACTS AND LOCATIONS:
Overall Officials: Hege Ihle-Hansen, MD, Principal Investigator — Sykehuset Asker og Baerum
Locations (1):
- Sykehuset Asker og Baerum HF, Pb 83, 1309, Norway

REFERENCES:
- [Derived] Hagberg G, Ihle-Hansen H, Fure B, Thommessen B, Ihle-Hansen H, Oksengard AR, Beyer MK, Wyller TB, Muller EG, Pendlebury ST, Selnes P. No evidence for amyloid pathology as a key mediator of neurodegeneration post-stroke - a seven-year follow-up study. BMC Neurol. 2020 May 8;20(1):174. doi: 10.1186/s12883-020-01753-w. PMID 32384876
- [Derived] Ihle-Hansen H, Hagberg G, Fure B, Thommessen B, Fagerland MW, Oksengard AR, Engedal K, Selnes P. Association between total-Tau and brain atrophy one year after first-ever stroke. BMC Neurol. 2017 Jun 5;17(1):107. doi: 10.1186/s12883-017-0890-6. PMID 28583116
- [Derived] Ihle-Hansen H, Thommessen B, Fagerland MW, Oksengard AR, Wyller TB, Engedal K, Fure B. Blood pressure control to prevent decline in cognition after stroke. Vasc Health Risk Manag. 2015 Jun 9;11:311-6. doi: 10.2147/VHRM.S82839. eCollection 2015. PMID 26089677
- [Derived] Ihle-Hansen H, Thommessen B, Fagerland MW, Oksengard AR, Wyller TB, Engedal K, Fure B. Effect on anxiety and depression of a multifactorial risk factor intervention program after stroke and TIA: a randomized controlled trial. Aging Ment Health. 2014 Jul;18(5):540-6. doi: 10.1080/13607863.2013.824406. Epub 2013 Aug 20. PMID 23957255